CLINICAL TRIAL: NCT07142525
Title: Aesthetic and Functional Outcomes Following Hybrid Osteoplasty Versus Traditional Osteotomy in Rhinoplasty: A Randomized Controlled Trial
Brief Title: Hybrid Osteoplasty Versus Osteotomy in Rhinoplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Goran Latif Omer, Associate Professor, University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No. 159 (August 17th, 2025)
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Rhinoplasty Techniques
Keywords: Osteoplasty; Dorsal Hump; Rhinoplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid Osteoplasty (Experimental): Participants undergo dorsal hump reduction using a surgical burr (drill) without traditional dorsal osteotomy. The technique allows controlled bone contouring under direct visualization.
  Interventions: Procedure: Hybrid Osteoplasty
- Traditional Osteotomy and Rasping (Active Comparator): Participants undergo dorsal hump reduction using the conventional method of osteotomy combined with rasping. This is the established standard approach for contouring the nasal dorsum.
  Interventions: Procedure: Traditional Osteotomy and Rasping

INTERVENTIONS:
Procedure: Hybrid Osteoplasty — Open rhinoplasty with dorsal hump reduction performed using a powered surgical burr under irrigation and direct visualization. Bone is contoured gradually to achieve a smooth dorsum while preserving the keystone area. No dorsal osteotomy is performed in this arm. Cartilaginous work and adjunctive steps (e.g., septoplasty or tip refinement) are performed as clinically indicated but are not part of the intervention being tested.
  Other Names: Drill-Assisted Dorsal Hump Reduction; Power-Assisted Osteoplasty; Burr Osteoplasty
  Arms: Hybrid Osteoplasty
Procedure: Traditional Osteotomy and Rasping — Open rhinoplasty using the conventional technique for dorsal hump reduction. The bony hump is resected with a straight osteotome, followed by manual rasping to refine the nasal dorsum, with preservation of the keystone area. Powered burrs are not used for primary dorsal contouring in this arm. Cartilaginous work and adjunctive procedures may be performed as clinically indicated but are not part of the tested intervention.
  Other Names: Osteotome + Rasp Technique; Conventional Dorsal Hump Reduction
  Arms: Traditional Osteotomy and Rasping

SUMMARY:
This study is designed to compare two common techniques for reducing the nasal hump during rhinoplasty: the traditional method using osteotomes and rasps, and a newer technique called hybrid osteoplasty that uses a surgical drill. Both approaches aim to improve the appearance and function of the nose. The trial will measure pain, swelling, bruising, and the smoothness of the nasal bridge, as well as patient satisfaction and breathing outcomes. Participants will be followed for one year to assess both early healing and long-term results.

DETAILED DESCRIPTION:
This prospective randomized controlled trial will evaluate the aesthetic and functional outcomes of hybrid osteoplasty using a surgical burr compared with traditional osteotomy and rasping in primary open rhinoplasty patients presenting with dorsal humps. The study population consists of adults without prior nasal surgery, trauma, or congenital deformities. Patients are randomized into two groups: Group A (hybrid osteoplasty) and Group B (traditional osteotomy plus rasping).

The primary objective is to assess differences in postoperative pain, edema, ecchymosis, dorsal smoothness, contour regularity, and patient satisfaction. Secondary outcomes include functional improvement measured by the Nasal Obstruction Symptom Evaluation (NOSE) score, aesthetic satisfaction assessed by the Rhinoplasty Outcome Evaluation (ROE), and the rate of revision surgery within 12 months.

Follow-up assessments are scheduled on postoperative Days 1, 2, and 7, and at 1, 3, 6, and 12 months. Standardized photographic documentation will support aesthetic evaluation, while clinical scoring systems will provide objective and subjective outcome data. The trial is powered to identify whether hybrid osteoplasty offers advantages in contour refinement and reduced soft tissue trauma compared with conventional osteotomy-based approaches.

ELIGIBILITY:
Inclusion Criteria:

* Primary open rhinoplasty planned.
* Dorsal hump with bony or mixed component suitable for either technique.
* No prior nasal surgery or significant nasal trauma affecting dorsum.
* ASA I-III and fit for general anesthesia.
* Willing to provide written informed consent, including standardized photography.
* Able and willing to attend all follow-up visits through 12 months.

Exclusion Criteria:

* Revision rhinoplasty or prior osteotomy/osseocartilaginous work.
* Active infection, open lesions, or uncontrolled dermatologic conditions at operative field.
* Bleeding diathesis, platelet disorder, INR elevation, or anticoagulant/antiplatelet therapy that cannot be paused.
* Uncontrolled systemic disease (e.g., hypertension, diabetes) or ASA ≥ IV.
* Pregnancy or breastfeeding.
* Chronic isotretinoin use within past 6 months or long-term systemic corticosteroid use.
* Concurrent interventional study that may affect healing or outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Rhinoplasty Outcome Evaluation (ROE) Score from Baseline to 12 Months | Baseline (preoperative) and 12 months post-operation.
  ROE (Rhinoplasty Outcome Evaluation) questionnaire scored 0-100 (higher = greater satisfaction). Score calculated per instrument guidance from the 6 items, converted to 0-100. Change is 12-month minus preoperative score.
Mean Dorsal Contour Irregularity Score on Blinded Photographic Assessment at 12 Months | 12 months post-operation.
  Standardized 7-view photographs rated by three blinded surgeons using a 4-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe irregularity). Primary analysis compares group means; inter-rater agreement assessed.
Mean Periorbital Edema Score on 4-Point Clinician Scale at Day 1 and Day 7 | Post-op Day 1 and Day 7.
  3 Clinicians-rated 4-point edema scale (0 = none, 1 = mild, 2 = moderate, 3 = severe).
Mean Periorbital Ecchymosis Score on 4-Point Clinician Scale at Day 1 and Day 7 | Post-op Day 1 and Day 7.
  3 Clinician-rated 4-point ecchymosis scale (0-3).
Proportion of Participants with Residual Hump or Dorsal Depression on Blinded Photographic Assessment at 12 Months | 12 months post-operation
  Blinded photographic assessment for remnant hump or depression (present/absent), by 3 assessors.
Proportion of Participants with Nasal Dorsum Width Symmetry at 12 Months | 12 months post-operation
  Symmetry rated by 3 blinded assessors on 3-point scale (symmetric / mildly asymmetric / asymmetric)
Number of Participants Requiring Unplanned Revision Surgery within 12 Months | Within 12 months post-operation
  Any unplanned surgical revision related to the nasal dorsum

SECONDARY OUTCOMES:
Proportion of Participants with Smooth Nasal Dorsum (Non-Blinded Binary Assessment) at 12 Months | 12 months post-operation
  Smooth vs Irregular, reported by 3 assessors
Mean Change in Nasal Obstruction Symptom Evaluation (NOSE) Score from Baseline to 12 Months | Baseline (preoperative) and 12 months post-operation.
  NOSE questionnaire scored 0-100 (higher = worse obstruction). Change is 12-month minus preoperative score; negative values indicate improvement.
Mean Pain Score on 0-10 Visual Analogue Scale at Post-Op Day 0 and Day 7 | Post-op Day 0 and Day 7
  Pain measured on a 0-10 visual analogue scale (higher = more pain)
Proportion of Participants with Palpable or Visible Dorsal Callus on Clinical Exam at 3 and 6 Months | 3 and 6 months post-operation
  Presence of palpable or visible dorsal callus on clinical exam (Yes/No). 3 assessors.

CONTACTS AND LOCATIONS:
Overall Officials: Goran L Omer, PhD, Study Chair — University of Sulaimani
Locations (1):
- Royal Hospital, Sulaymaniyah, KRI, Iraq

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results will be shared, including baseline demographic information, surgical technique allocation, intraoperative variables, and postoperative outcome measures (pain scores, edema, ecchymosis, ROE scores, NOSE scores, blinded photographic assessments, and revision status). Data will be available in de-identified form upon reasonable request to the principal investigator after publication of the primary results. Supporting documents, including the study protocol and statistical analysis plan, will also be made available.
Time Frame: IPD and supporting information will be available beginning after publication of the primary study results and will remain available for a minimum of 5 years thereafter.
Access Criteria: De-identified IPD and supporting documents will be made available to qualified researchers affiliated with academic institutions or recognized research organizations. Requests must include a methodologically sound proposal and will be reviewed by the principal investigator. Approved requestors will be required to sign a data use agreement ensuring compliance with ethical and confidentiality standards. Data will be provided in de-identified format via secure transfer.

REFERENCES:
- [Background] Azizli E, Bayar Muluk N, Dundar R, Cingi C. A new preservation technique for dehumping the dorsum. Eur Rev Med Pharmacol Sci. 2023 Mar;27(2 Suppl):57-62. doi: 10.26355/eurrev_202303_31703. PMID 36971222
- [Background] Ferreira MG, Monteiro D, Reis C, Almeida e Sousa C. Spare Roof Technique: A Middle Third New Technique. Facial Plast Surg. 2016 Feb;32(1):111-6. doi: 10.1055/s-0035-1570503. Epub 2016 Feb 10. PMID 26862972
- [Background] Aldosari BF, Alhajress RI, Bogari AO. Hump Rasping Using Powered Instruments: A Retrospective Review. Plast Reconstr Surg Glob Open. 2024 Sep 10;12(9):e6153. doi: 10.1097/GOX.0000000000006153. eCollection 2024 Sep. PMID 39258281
- [Background] Lal GN, Ghosh P. Use of drill in rhinoplasty (a case report). Indian J Otolaryngol Head Neck Surg. 1999 Jan;51(1):90-2. doi: 10.1007/BF02996859. PMID 23119498
- [Background] Goodman WS. The rotating burr in rhinoplasty. Arch Otolaryngol. 1981 Jul;107(7):436-8. doi: 10.1001/archotol.1981.00790430038010. No abstract available. PMID 7247809
- [Background] Avashia YJ, Marshall AP, Allori AC, Rohrich RJ, Marcus JR. Decision-Making in Middle Vault Reconstruction following Dorsal Hump Reduction in Primary Rhinoplasty. Plast Reconstr Surg. 2020 Jun;145(6):1389-1401. doi: 10.1097/PRS.0000000000006850. PMID 32195860
- [Background] Barrett DM, Casanueva F, Wang T. Understanding Approaches to the Dorsal Hump. Facial Plast Surg. 2017 Apr;33(2):125-132. doi: 10.1055/s-0037-1598033. Epub 2017 Apr 7. PMID 28388791
- [Background] Fuller JC, Hilger PA. Modified Skoog Method for Hump Reduction. Facial Plast Surg Clin North Am. 2021 Feb;29(1):131-139. doi: 10.1016/j.fsc.2020.09.008. PMID 33220838
- [Background] Sowder JC, Thomas AJ, Gonzalez CD, Limaye NS, Ward PD. Use of Spreader Flaps Without Dorsal Hump Reduction and the Effect on Nasal Function. JAMA Facial Plast Surg. 2017 Jul 1;19(4):287-292. doi: 10.1001/jamafacial.2016.2057. PMID 28241228
- [Background] Azizzadeh B, Reilly M. Dorsal Hump Reduction and Osteotomies. Clin Plast Surg. 2016 Jan;43(1):47-58. doi: 10.1016/j.cps.2015.09.022. Epub 2015 Oct 23. PMID 26616694
- [Background] Roostaeian J, Unger JG, Lee MR, Geissler P, Rohrich RJ. Reconstitution of the nasal dorsum following component dorsal reduction in primary rhinoplasty. Plast Reconstr Surg. 2014 Mar;133(3):509-518. doi: 10.1097/01.prs.0000438453.29980.36. PMID 24263393
- [Background] Rohrich RJ, Muzaffar AR, Janis JE. Component dorsal hump reduction: the importance of maintaining dorsal aesthetic lines in rhinoplasty. Plast Reconstr Surg. 2004 Oct;114(5):1298-308; discussion 1309-12. doi: 10.1097/01.prs.0000135861.45986.cf. PMID 15457053